CLINICAL TRIAL: NCT05848622
Title: Gait Rehabilitation to Treat FastOA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Arthritis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 21-1489b
Record Dates: First submitted 2023-04-14; First posted 2023-05-08 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Anterior Cruciate Ligament Injuries; Post-traumatic Osteoarthritis; Knee Osteoarthritis; Osteo Arthritis Knee; Knee Injuries; Cartilage, Articular; Gait
Keywords: Biofeedback; FastOA
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Osteoarthritis, Knee; Knee Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real-time gait biofeedback (RTGBF) (Active Comparator): The RTGBF regimen delivers biofeedback that cues a personalized target to normalize vertical ground reaction force (vGRF) of each limb.
  Interventions: Behavioral: Real-time gait biofeedback
- Sham real-time gait biofeedback (Sham RTGBF) (Sham Comparator): The Sham RTGBF regimen will receive biofeedback that cues their habitual step length determined during the accommodation period on the first session of treadmill walking.
  Interventions: Behavioral: Sham real-time gait biofeedback

INTERVENTIONS:
Behavioral: Real-time gait biofeedback — The RTGBF interventions will include eighteen step gait training sessions. The intervention will gradually increase to 3,000 steps at the 5th session with 100% feedback. During the remaining sessions, the intervention will include 3,000 steps, but the feedback will be gradually tapered off starting with the 11th session.
  Arms: Real-time gait biofeedback (RTGBF)
Behavioral: Sham real-time gait biofeedback — The Sham RTGBF interventions will include eighteen step gait training sessions. The intervention will gradually increase to 3,000 steps at the 5th session with 100% feedback. During the remaining sessions, the intervention will include 3,000 steps, but the feedback will be gradually tapered off starting with the 11th session.
  Arms: Sham real-time gait biofeedback (Sham RTGBF)

SUMMARY:
The purpose of this study is to determine the effects of real-time gait biofeedback delivered over a 6-week period on early markers of FastOA and conduct 6-week and 6-month follow-up assessments in anterior cruciate ligament reconstructed patients.

ELIGIBILITY:
Inclusion Criteria:

* Have completed all other formal physical therapy
* Are between the ages of 16 and 35
* Underwent an anterior cruciate ligament reconstruction (ACLR) between 6 and 60 months prior to enrollment
* Demonstrate underloading during gait (vGRF- impact peak <1.12 x BW)

Exclusion Criteria:

* A multiple ligament surgery (i.e., PCL)
* A lower extremity fracture (i.e., displaced tibial plateau fracture)
* Knee osteoarthritis
* The participant has a BMI ≥ 36.

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-06-13 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Mean Change from Baseline to Week 6 in Vertical Ground Reaction Force | Baseline, Week 6
  Participants walk on a dual-belt force-sensing treadmill for 3000 steps while vertical ground reaction forces are collected. Change score (Post-Pre) loading rate calculated as the peak of the first time derivative of the vertical ground reaction force time series curve during the first 50% of the stance phase. This will be collected at Baseline (pre-intervention) and 6 weeks posttest. An increase in vertical ground reaction force at 6 weeks from baseline indicates improved gait mechanics.
Mean Change from Baseline to Month 6 in Vertical Ground Reaction Force | Baseline, Month 6
  Participants walk on a dual-belt force-sensing treadmill for 3000 steps while vertical ground reaction forces are collected. Change score (Post-Pre) loading rate calculated as the peak of the first time derivative of the vertical ground reaction force time series curve during the first 50% of the stance phase. This will be collected at Baseline (pre-intervention) and 6 months posttest. An increase in vertical ground reaction force at 6 months from baseline indicates improved gait mechanics.
Mean Change from Baseline to Week 6 in Knee Joint Contact Forces | Baseline, Week 6
  Participants walked on a dual-belt force-sensing treadmill for 3000 steps while lower limb kinematics and kinetics were collected. Walking kinematics and kinetics are submitted to musculoskeletal modeling simulations used to determine the magnitude and location of knee joint contact forces. Change score (post-pre) joint contact forces during the first 50% of the stance phase will be calculated. This will be collected at Baseline (pre-intervention) and 6 weeks posttest. An increase in vertical ground reaction force at 6 weeks from baseline indicates improved gait mechanics.
Mean Change from Baseline to Month 6 in Knee Joint Contact Forces | Baseline, Month 6
  Participants walked on a dual-belt force-sensing treadmill for 3000 steps while lower limb kinematics and kinetics were collected. Walking kinematics and kinetics are submitted to musculoskeletal modeling simulations used to determine the magnitude and location of knee joint contact forces. Change score (post-pre) joint contact forces during the first 50% of the stance phase will be calculated. This will be collected at Baseline (pre-intervention) and 6 months posttest. An increase in vertical ground reaction force at 6 months from baseline indicates improved gait mechanics.
Mean Change from Baseline to Week 6 in Tibial Cartilage Strain | Baseline, Week 6
  MRI imaging provided measures of tibial cartilage thickness before and after a standardized walking protocol that were used to measure cartilage strain. The articular cartilage is viscoelastic, and cartilage strain refers to the deformation profiles of the articular cartilage after applying a load. This will be collected at Baseline (pre-intervention) and 6 weeks posttest. More defuse cartilage strain across the knee joint reflects a better outcome.
Mean Change from Baseline to Month 6 in Tibial Cartilage Strain | Baseline, Month 6
  MRI imaging provided measures of tibial cartilage thickness before and after a standardized walking protocol that were used to measure cartilage strain. The articular cartilage is viscoelastic, and cartilage strain refers to the deformation profiles of the articular cartilage after applying a load. This will be collected at Baseline (pre-intervention) and 6 months posttest. More defuse cartilage strain across the knee joint reflects a better outcome.
Mean Change from Baseline to Week 6 in the Knee Injury and Osteoarthritis Outcome Quality of Life Subscale Score | Baseline, Week 6
  Knee injury Osteoarthritis Outcome Score (KOOS) Quality of Life subscale to measure knee-related quality of life at pre-intervention (baseline). This will be collected at Baseline (pre-intervention) and 6 weeks posttest. A higher score indicates better knee-related quality of life. Range: 0-100.
Mean Change from Baseline to Month 6 in the Knee Injury and Osteoarthritis Outcome Quality of Life Subscale Score | Baseline, Month 6
  Knee injury Osteoarthritis Outcome Score (KOOS) Quality of Life subscale to measure knee-related quality of life at pre-intervention (baseline). This will be collected at Baseline (pre-intervention) and 6 months posttest. A higher score indicates better knee-related quality of life. Range: 0-100.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing Biomarker Chemokine (Monocyte Chemoattractant Protein-1 (MCP-1)). | Baseline, Week 6
  Blood for serum-based biomarker chemokine (monocyte chemoattractant protein-1 (MCP-1)). This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing Biomarker Chemokine (Monocyte Chemoattractant Protein-1 (MCP-1)). | Baseline, Month 6
  Blood for serum-based biomarker chemokine (monocyte chemoattractant protein-1 (MCP-1)). This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing Degenerative Matrix Metalloproteinase-1 (MMP-1) Enzyme | Baseline, Week 6
  Blood for serum-based biomarker degenerative matrix metalloproteinase-1 (MMP-1) enzyme. This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing Degenerative Matrix Metalloproteinase-1 (MMP-1) Enzyme | Baseline, Month 6
  Blood for serum-based biomarker degenerative matrix metalloproteinase-1 (MMP-1) enzyme. This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing Degenerative Matrix Metalloproteinase-3 (MMP-3) Enzyme | Baseline, Week 6
  Blood for serum-based biomarker degenerative matrix metalloproteinase-3 (MMP-3) enzyme. This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing Degenerative Matrix Metalloproteinase-3 (MMP-3) Enzyme | Baseline, Month 6
  Blood for serum-based biomarker degenerative matrix metalloproteinase-3 (MMP-3) enzyme. This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing Degenerative Matrix Metalloproteinase-9 (MMP-9) Enzyme | Baseline, Week 6
  Blood for serum-based biomarker degenerative matrix metalloproteinase-9 (MMP-9) enzyme. This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing Degenerative Matrix Metalloproteinase-9 (MMP-9) Enzyme | Baseline, Month 6
  Blood for serum-based biomarker degenerative matrix metalloproteinase-9 (MMP-9) enzyme. This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing the Inflammatory Response via Interleukin 6 (IL-6) | Baseline, Week 6
  Blood for serum-based biomarker interleukin 6 (IL-6). This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing the Inflammatory Response via Interleukin 6 (IL-6) | Baseline, Month 6
  Blood for serum-based biomarker interleukin 6 (IL-6). This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing Tumor Necrosis Factor Alpha (TNF-Alpha) | Baseline, Week 6
  Blood for serum-based biomarker Tumor Necrosis Factor Alpha (TNF-Alpha). This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing Tumor Necrosis Factor Alpha (TNF-Alpha) | Baseline, Month 6
  Blood for serum-based biomarker Tumor Necrosis Factor Alpha (TNF-Alpha). This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing a Disintegrin and Metalloproteinase with thrombospondin Motifs-4 (ADAMTS-4) | Baseline, Week 6
  Blood for serum-based biomarker a disintegrin and metalloproteinase with thrombospondin motifs-4 (ADAMTS-4). This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing a Disintegrin and Metalloproteinase with thrombospondin Motifs-4 (ADAMTS-4) | Baseline, Month 6
  Blood for serum-based biomarker a disintegrin and metalloproteinase with thrombospondin motifs-4 (ADAMTS-4). This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing a Marker of Cartilage Turnover (Cartilage Oligomeric Matrix Protein (COMP)) | Baseline, Week 6
  Blood for serum-based biomarker marker of cartilage turnover (cartilage oligomeric matrix protein (COMP)). This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing a Marker of Cartilage Turnover (Cartilage Oligomeric Matrix Protein (COMP)) | Baseline, Month 6
  Blood for serum-based biomarker marker of cartilage turnover (cartilage oligomeric matrix protein (COMP)). This will be collected at Baseline (pre-intervention) and 6 months posttest.
Mean Change from Baseline to Week 6 in Joint Tissues Metabolism by Assessing a Marker of Cartilage Turnover C-Terminal Crosslinked Telopeptide-II (CTXII) | Baseline, Week 6
  Urine for urine-based biomarker marker of cartilage degradation C-terminal crosslinked telopeptide-II (CTXII). This will be collected at Baseline (pre-intervention) and 6 weeks posttest.
Mean Change from Baseline to Month 6 in Joint Tissues Metabolism by Assessing a Marker of Cartilage Turnover C-Terminal Crosslinked Telopeptide-II (CTXII) | Baseline, Month 6
  Urine for urine-based biomarker marker of cartilage degradation C-terminal crosslinked telopeptide-II (CTXII). This will be collected at Baseline (pre-intervention) and 6 months posttest.

SECONDARY OUTCOMES:
Change in the International Knee Documentation Committee Subjective Knee Evaluation Form Score | Up to 6 months
  The International Knee Documentation Committee (IKDC) Subjective Knee Evaluation form is a 10-item survey that determines patient-reported knee-related function. This will be collected at Baseline (pre-intervention), 6-week posttest, and 6-month posttest. A higher score indicates better knee function. Range: 0-100.
Change in the Tegner Activity Scale Score | Up to 6 months
  The Tegner Activity Scale (TAS) to quantify activity levels in individuals with ACL injury on an 11-point Likert scale. A higher score indicates a higher level of activity (e.g., a 10 indicates participants compete in professional or collegiate levels of sport on a regular basis while a 0 indicates indicates that participants are unable to complete any sport or recreational activity due to disability). This will be collected at Baseline (pre-intervention), 6-week posttest, and 6-month posttest.
Change in the Anterior Cruciate Ligament Return to Sport After Injury Scale Score | Up to 6 months
  The Anterior Cruciate Ligament Return to Sport After Injury (ACL-RSI) scale to measure an individual's psychological readiness to return to sport. Range: 0-100 points. A lower score on this questionnaire indicates poorer psychological readiness. This will be collected at Baseline (pre-intervention), 6-week posttest, and 6-month posttest.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pietrosimone, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB and an executed data use/sharing agreement with UNC.